CLINICAL TRIAL: NCT03378661
Title: Phase 2 Randomized, Multicenter, Safety and Efficacy Trial to Evaluate Different Oral Benznidazole Monotherapy and Benznidazole/E1224 Combination Regimens for the Treatment of Adult Patients With Chronic Indeterminate Chagas Disease
Brief Title: BENDITA BEnznidazole New Doses Improved Treatment and Associations
Acronym: BENDITA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Drugs for Neglected Diseases (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DNDi-CH-E1224-003
Record Dates: First submitted 2017-11-23; First posted 2017-12-20 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Chagas Disease
Keywords: Chronic, Indeterminate
MeSH Terms: conditions — Chagas Disease; Bronchiolitis Obliterans Syndrome | interventions — benzonidazole; fosravuconazole L-lysine ethanolate; Prodrugs

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Dummy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- BZN STD Regimen (Experimental): Benznidazole (100 mg and 50 mg) tablets by mouth, every 12 hours for 8 weeks.
  Three E1224 Placebo 100 mg capsules by mouth, everyday on days 1 to 3, followed by three E1224 Placebo 100 mg capsules by mouth, once weekly (starting on week 2) for 7 weeks.
  Interventions: Drug: Benznidazole; Drug: E1224 Placebo
- BZN 300 mg - 4 wks (Experimental): Benznidazole (100 mg and 50 mg) tablets by mouth, every 12 hours for 4 weeks, followed by:
  Benznidazole Placebo (100 mg and 50 mg) tablets by mouth, every 12 hours for 4 weeks.
  Three E1224 Placebo 100 mg capsules by mouth, everyday on days 1 to 3, followed by three E1224 Placebo 100 mg capsules by mouth, once weekly (starting on week 2) for 7 weeks.
  Interventions: Drug: Benznidazole; Drug: E1224 Placebo; Drug: Benznidazole Placebo
- BZN 300 mg - 2 wks (Experimental): Benznidazole (100 mg and 50 mg) tablets by mouth, every 12 hours for 2 weeks, followed by:
  Benznidazole Placebo (100 mg and 50 mg) tablets by mouth, every 12 hours for 6 weeks.
  Three E1224 Placebo 100 mg capsules by mouth, everyday on days 1 to 3, followed by three E1224 Placebo 100 mg capsules by mouth, once weekly (starting on week 2) for 7 weeks.
  Interventions: Drug: Benznidazole; Drug: E1224 Placebo; Drug: Benznidazole Placebo
- BZN 150 mg - 4 wks (Experimental): Benznidazole (100 mg and 50 mg) tablets and Benznidazole Placebo (100 mg and 50 mg) tablets by mouth, in two separate daily doses for 4 weeks, followed by:
  Benznidazole Placebo (100 mg and 50 mg) tablets by mouth, every 12 hours for 4 weeks.
  Three E1224 Placebo 100 mg capsules by mouth, everyday on days 1 to 3, followed by three E1224 Placebo 100 mg capsules by mouth, once weekly (starting on week 2) for 7 weeks.
  Interventions: Drug: Benznidazole; Drug: E1224 Placebo; Drug: Benznidazole Placebo
- BZN 150 mg - 4 wks / E1224 300 mg (Experimental): Benznidazole (100 mg and 50 mg) tablets and Benznidazole Placebo (100 mg and 50 mg) tablets by mouth, in two separate daily doses for 4 weeks, followed by:
  Benznidazole Placebo (100 mg and 50 mg) tablets by mouth, every 12 hours for 4 weeks.
  Three E1224 100 mg capsules by mouth, everyday on days 1 to 3, followed by three E1224 100 mg capsules by mouth, once weekly (starting on week 2) for 7 weeks. (total dose: 3000 mg).
  Interventions: Drug: Benznidazole; Drug: E1224; Drug: Benznidazole Placebo
- BZN 300 mg (weekly) 8 wks / E1224 300 mg (Experimental): Benznidazole (100 mg and 50 mg) tablets by mouth, once weekly for 8 weeks (total 8 days of intermittent treatment) and Benznidazole Placebo (100 mg and 50 mg) tablets by mouth, in the other 6 days of the week for 8 weeks
  Three E1224 100 mg capsules by mouth, everyday on days 1 to 3, followed by three E1224 100 mg capsules by mouth, once weekly (starting on week 2) for 7 weeks. (total dose: 3000 mg).
  Interventions: Drug: Benznidazole; Drug: E1224; Drug: Benznidazole Placebo
- Placebo (Placebo Comparator): Benznidazole Placebo (100 mg and 50mg) tablets by mouth, every 12 hours for 8 weeks.
  Three E1224 Placebo 100 mg capsules by mouth, everyday on days 1 to 3, followed by three E1224 Placebo 100 mg capsules by mouth, once weekly (starting on week 2) for 7 weeks.
  Interventions: Drug: E1224 Placebo; Drug: Benznidazole Placebo

INTERVENTIONS:
Drug: Benznidazole — Benznidazole tablet
  Other Names: Abarax®; N-benzil-2-nitro-1-imidazolacetamide); Lafepe Benznidazol; ABALEA®
  Arms: BZN 150 mg - 4 wks; BZN 150 mg - 4 wks / E1224 300 mg; BZN 300 mg (weekly) 8 wks / E1224 300 mg; BZN 300 mg - 2 wks; BZN 300 mg - 4 wks; BZN STD Regimen
Drug: E1224 — E1224 capsules
  Other Names: Fosravuconazole; E1224 (prodrug for active ingredient Ravuconazole)
  Arms: BZN 150 mg - 4 wks / E1224 300 mg; BZN 300 mg (weekly) 8 wks / E1224 300 mg
Drug: E1224 Placebo — E1224 matched placebo capsules
  Other Names: Placebo (for E1224)
  Arms: BZN 150 mg - 4 wks; BZN 300 mg - 2 wks; BZN 300 mg - 4 wks; BZN STD Regimen; Placebo
Drug: Benznidazole Placebo — Benznidazole matched placebo tablets
  Other Names: Placebo (for Benznidazole)
  Arms: BZN 150 mg - 4 wks; BZN 150 mg - 4 wks / E1224 300 mg; BZN 300 mg (weekly) 8 wks / E1224 300 mg; BZN 300 mg - 2 wks; BZN 300 mg - 4 wks; Placebo

SUMMARY:
Recent scientific advances have provided further impetus to develop new therapeutic approaches for Chagas Disease (CD) using different doses and duration of BZN, as well as combinations directed at multiple therapeutic targets to improve treatment response and tolerability and reduce the potential for development of resistance.

This project focuses on the proof-of-concept evaluation of improved treatment regimens of BZN, with the assessment of new BZN-sparing regimens in monotherapy and in combination with E1224.

DETAILED DESCRIPTION:
The current treatment for Chagas disease has significant limitations, including long treatment durations, safety and tolerability concerns and is currently limited to two nitro-heterocyclic drugs, nifurtimox and benznidazole (BZN). BZN, a nitroimidazole introduced by Roche in 1971, is marketed by Laboratório Farmacêutico do Estado de Pernambuco S/A - LAFEPE and Laboratorio ELEA - Argentina. It is supplied in tablets strengths of 12.5, 50 and 100 mg, administered twice daily at a dose of 5 mg/kg body weight/day for adults and 5-10 mg/kg body weight/day for children for 30-60 days. Notably, the current regimens with BZN for the treatment of adults with CD likely represent the maximum dosing case scenario in terms of dose, duration and schedule of administration (Chagas expert meeting DNDi. January 2014. GVA).

Doses and duration of treatment for CD have not been evaluated systematically. Current treatment regimens and dosing intervals have been derived from decades-old patient series and with very limited direct comparisons. Data from recently concluded trials suggest existing opportunities for optimisation of the treatment regimens of BZN.

A (Drugs for Neglected Disease initiative) DNDi-sponsored Phase 2, proof-of-concept clinical trial on E1224 and Benznidazole (BZN) in adults with chronic indeterminate CD, conducted between 2011 and 2013 in Bolivia, showed that all BZN-treated patients had cleared parasite DNA after 2 weeks of treatment and 81% sustained the parasite clearance at 12 months after treatment. At end-of treatment (EOT, Day 65), E1224 was found to be efficacious in clearing T. cruzi parasites when compared to placebo. However, at 12 months less than one third of patients sustained parasite clearance. The trial safety data also indicated a proportion of patients (10-20%) who do not complete treatment in conditions of use, the majority due to adverse drug reactions (ADRs) and the long treatment duration.

Taking into consideration the efficacy gap with about 80% sustained response and a tolerability gap, with a proportion of patients (10-20%) who do not complete treatment, two approaches for Chagas treatment optimization are to be pursued:

1. A change in the current adult dosing regimen for BNZ to reduce exposure and improve tolerability while maintaining efficacy; and
2. The development of a combination therapy to improve efficacy while maintaining or improving tolerability. The combination therapy aims to address the efficacy gap and may or may not address tolerability gap.

With regards to the dosing regimen, population-pharmacokinetics studies observed BZN plasma concentrations in children were significantly lower than those previously reported in adults (treated with comparable mg/kg doses). At the same time, all children had parasite clearance, few adverse reactions to the drug. Recent population PK data in adults suggested that the current BZN dosing regimen (2.5 mg/kg/12 h) may lead to overexposure in the majority of patients. Dosing simulations suggested that a BNZ dose of 2.5 mg/kg/24 h would adequately keep BNZ trough plasma concentrations within the recommended target range for the majority of patients. There are also opportunities for evaluation of fixed dose regimens for adult dosing, rather than mg/kg calculations, with increased ease-of-use and potential for improved compliance in scaling up treatment of CD. Intermittent dosing regimens was also evaluated in murine model of chronic CD and in a pilot follow-up trial with 17 adult patients with chronic CD was, with similar parasitological cure rates to standard treatment.

Likewise, several controlled observational trials with BZN, 5 mg/kg/day for 30 or 60 days have shown a reduction in the progression of heart disease serological and sero-negative conversion up to 60% in children and 30% in adults. Different publications showed anti-parasitic efficacy of treatment regimens with 30 and 60 days, and of incomplete treatment of 10 days. Combination therapy is a well-recognized treatment modality in many disease settings, including cancer, cardiovascular disease, and infectious diseases. Several infectious diseases such as tuberculosis, malaria, leprosy, and AIDS only came under control and were effectively treated after introduction of combinations of drugs that utilize different mechanisms of action.

E1224 is a water-soluble monolysine salt form of the ravuconazole (RAV) pro-drug (which is a phosphonooxymethyl ether derivative of RAV). It is a broad-spectrum triazole antifungal.

Pooled safety data for the monolysine prodrug E1224 from Phase 1 and 2 trials indicated that E1224 was generally well tolerated and exhibited a safety profile quite similar to other azoles. Adverse events occurring in greater than 3% of E1224 recipients, with a dose-dependent pattern and at rates higher than those observed in placebo recipients included nausea, abnormalities in liver enzymes, dizziness, anxiety, and contact dermatitis.

Safety evaluations indicated relatively mild, transient, and asymptomatic increases in liver enzymes - completely reversible upon discontinuation of therapy. Phase 1 cardiac safety evaluations showed that E1224 administration did not result in QTc interval prolongation.

Experimental data suggest a positive interaction between BZN and azole compounds for the treatment of Chagas disease.18 A Phase 1 drug-drug interaction trial was designed to assess the pharmacokinetics (PK) and safety interaction of BNZ and E1224 co-administered daily for a total of 54 days (Day 4 to Day 15- E1224 multiple dose 400 mg loading dose once daily for 3 days, followed by maintenance dose 100mg once daily for 9 days (from Day 7 to Day 15); Day 9 BNZ single dose (2.5 mg/kg); and Day 12 to Day 15 BNZ multiple dose (2.5 mg/kg twice daily)). The trial was conducted in Argentina and was concluded in early 2015, with enrolment of 28 healthy male volunteers. Both compounds were well tolerated, in monotherapy and combination. There were no treatment discontinuations or serious adverse events. Transient, minor, non-concomitant increase in bilirubin and liver transaminases occurred in 2 patients in a pattern not suggestive of drug effect. There was no interaction of RAV on BNZ PK and the limited impact of BNZ on RAV PK, suggesting that co-administration of RAV and BNZ may not require any E1224 dosing adaptation. The lack of clinically relevant safety findings provided support for follow-up evaluation of the two compounds in combination.

In conclusion, recent scientific advances have provided further impetus to develop new therapeutic approaches for CD using different doses and duration of BZN, as well as combinations directed at multiple therapeutic targets to improve treatment response and tolerability and reduce the potential for development of resistance.

This project focuses on the proof-of-concept evaluation of improved treatment regimens of BZN, with the assessment of new BZN-sparing regimens in monotherapy and in combination with E1224.

ELIGIBILITY:
Screening criteria

* Signed, written informed consent form
* Age >18 to <50 years
* Weight >50 kg to <80 kg
* Diagnosis of T. cruzi infection by: Conventional serology (a minimum of two positive tests [Conventional ELISA, Recombinant Elisa and/or Indirect Immunofluorescence (IIF)])
* Ability to comply with all protocol specified tests and visits and have a permanent address
* Patients must be residents of areas free of vectorial transmission (Triatoma infestans). For this protocol, it will be accepted the status of Vectorial Transmission Interruption or Consolidation as per the definition of PAHO/WHO, or the Local Health Program.
* No signs and/or symptoms of the chronic cardiac and/or digestive form of CD
* No acute or chronic health conditions, that in the opinion of the PI, may interfere with the efficacy and/or safety evaluation of the trial drug (such as acute infections, history of HIV infection, liver and renal disease requiring treatment)
* No formal contraindication to BZN (according to the Summary of Product Characteristics) and E1224 (according to the Investigator's Brochure) Note: The contraindications described for Benznidazole and E1224 are essentially hypersensitivity to the active ingredient or any excipient. In the case of hepatic or renal impairment or blood dyscrasia, the medication should only be administered under strict medical supervision. During all the treatment period, the blood count will be monitored, with special attention to leucocytes. Subjects will be indicated about the need of no alcohol intake.
* No history of hypersensitivity, allergic, or serious adverse reactions to any of the "azoles" compound, and/or its components
* No history of CD treatment with BZN or NFX at any time in the past
* No history of systemic treatment with itraconazole, ketoconazole, posaconazole, isavuconazole, or allopurinol in the past
* No history of alcohol abuse or any other drug addiction (as specified in the Study Manual of Operations)
* No condition that prevents patient from taking oral medication
* No concomitant or anticipated use of drugs that are either sensitive CYP3A4 substrates and/or extensively metabolized by CYP3A4 with a narrow therapeutic range (as per Appendix 2)
* No medical history of Familial Short QT syndrome or concomitant therapy with medications that can shorten the QT interval (as per Appendix 2)
* No family history of sudden death
* No family history of sudden infant death syndrome

Inclusion criteria

Following the screening period, patients must meet ALL of the following inclusion criteria to be eligible for randomization:

* Confirmed diagnosis of T. cruzi infection by: Serial qualitative PCR (three samples collected over a single day, at least one of which must be positive) AND Conventional serology (a minimum of two positive tests must be positive [Conventional ELISA, Recombinant Elisa and/or IIF)
* Women in reproductive age must have a negative serum pregnancy test at screening, must not be breastfeeding, and must use a double barrier method of contraception to avoid pregnancy throughout a clinical trial and for 3 months after completion of the trial, in such a manner that the risk of pregnancy is minimized especially during exposure to treatment. Women who are using oral, implanted, or injectable contraceptive hormones or mechanical products such as an intrauterine device with a hormonal component are required to use an additional barrier method of contraception for the time period specified.
* Normal EKG (PR ≤200 msec, QRS <120 msec, and QTc ≥350 msec and ≤450 msec interval durations in males and QTc ≤470 msec in women) at screening.

Exclusion criteria

The presence of any of the following will exclude a patient from trial randomization:

* Signs and/or symptoms of chronic cardiac and/or digestive form of CD
* History of cardiomyopathy, heart failure, or ventricular arrhythmia.
* History of digestive surgery or mega syndromes.
* Any other acute or chronic health conditions that, in the opinion of the PI, may interfere with the efficacy and/or safety evaluation of the trial drug (such as acute infections, history of HIV infection, diabetes, uncontrolled systolic/diastolic blood pressure, liver, and renal disease requiring medical treatment).
* Laboratory test values considered clinically significant or out of the allowable range at selection period as follows:
* Total WBC must be within the normal range, with an acceptable margin of +/- 5% (3,800 - 10,500/mm3).
* Platelets must be within the normal range up to 550,000/mm3
* Total bilirubin must be within the normal range
* Transaminases (ALT and AST) must be within the normal range, with an acceptable margin of 25% above the upper limit of normality (ULN), <1.25 x ULN.
* Creatinine must be within an acceptable margin of 10% above the ULN, <1.10 x ULN.
* Alkaline phosphatase must be within the normal range up to Grade 1 CTCAE (< 2.5 x ULN)
* GGT must be within the normal range up to 2x ULN.
* Fasting glucose must be within the normal range
* Electrolytes (Ca, Mg, K) must be within the normal range
* If the results of the blood tests (hematology and biochemistry) are out of the ranges defined above, but within the limits of CTCAE (version 4.03) Grade 1, and the laboratory finding is considered as non-clinically significant, a new sample can be collected for a retest. Only one retest will be allowed within the screening period.
* If the result of retest is within the margins defined above, the Investigator will review the parameter(s) together with all other medical information available (medical history, clinical examinations, vital signs, etc.) and upon his/her medical judgment will decide if the patient is eligible or not for trial randomization.
* Any condition that prevents the patient from taking oral medication
* Patients with history of allergy (serious or not), allergic skin rash, asthma, intolerance, sensitivity or photosensitivity to any drug
* Patients with any contra-indication (known hypersensitivity) to any nitroimidazoles, e.g. metronidazole.
* Any concomitant use of allopurinol, antimicrobial, or anti-parasitic agents.
* Any planned surgery likely to interfere with the trial conduction and/or treatment evaluation
* Unlikely to co-operate with the trial
* Any previous participation in any clinical trial for Chagas Disease treatment evaluation
* Participation in another trial at the same time or within 3 months prior to selection (according to local regulations)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2018-01-28 (Estimated); Study Completion 2018-07-27 (Estimated)

PRIMARY OUTCOMES:
Parasitological response as determined by serial negative qualitative PCR results (3 negative PCR results, from 3 samples to be collected in the same day) at EOT and sustained parasitological clearance until 6 months follow-up. | From the end of the treatment period up to 6 months.
  To determine the efficacy of different dosing regimens of orally administered BZN and BZN/E1224 in individuals with chronic indeterminate CD, by determining the proportion of patients who convert from positive to negative in serial, qualitative PCR test results (3 negative PCR results) at end of treatment (EOT) and sustain parasitological clearance at 6 months of follow-up, in comparison to placebo.
  For efficacy assessments, the EOT of each treatment arm will be defined in accordance to the duration of the treatment regimen. Sustained response will be assessed in all treatment arms using the same number of PCR samples (i.e., EOT; 12 weeks; 4 and 6 months).

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | Through study completion, i.e up to 12 months.
  The safety consists the description of each serious adverse event and adverse event (preferred term) per treatment group and classified by system organ. EkG and Laboratory abnormalities will be considered as Adverse Events.
Severity of Adverse Events (AEs) | Through study completion, i.e up to 12 months.
  The safety consists the description of each serious adverse event and adverse event (preferred term) per treatment group and classified by system organ. EkG and Laboratory abnormalities will be considered as Adverse Events.
Incidence of Serious Adverse Events (SAEs) and/or adverse events leading to treatment discontinuation | Through study completion, i.e up to 12 months
Sustained parasitological clearance at 12 weeks and 12 months of follow-up | From the end of the treatment period up to 12 months.
  To assess the sustained parasitological response at week 12 and 12 months for each of the regimens, in comparison with placebo.
  To determine the efficacy of the different dosing regimens in individuals with chronic indeterminate CD, by determining the proportion of patients who convert from positive to negative in serial, qualitative PCR test results (3 negative PCR results) at EOT, in comparison with placebo.
Parasite clearance as measured by qualitative PCR | Weeks 1, 2, 3, 4, 6, 10, 12, and at 4, 6, and 12 months follow-up
  To assess the time to parasite DNA clearance (below the Quantitative Polymerase Chain Reaction (qPCR) Limit of Detection (LOD) for each of the regimens.
  To assess the time to sustained clearance of parasitemia for each of the regimens.
Change in parasite load over time assessed as measured by quantitative PCR | Weeks 1, 2, 3, 4, 6, 10, 12, and at 4, 6, and 12 months follow-up.
  To measure the reduction in parasite load at weeks 1, 2, 3, 4, 6, 10, 12 and at 4, 6 and 12 months follow-up, as measured by quantitative PCR.
Serological response by conventional serology assessed at 12 months of follow up and non-conventional serology assessed at W12, 4, 6, and 12 months of follow up. (changes in titters over time) | From the end of the treatment period up to 12 months.
  To evaluate serological response by conventional serology at 12 months of follow up and non-conventional serology at week 12, 4, 6 and 12 months of follow up.

OTHER OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of ravuconazole and benznidazole | D0 (pre-dose), day 1 (post-dose), day 2, day 3, steady-state phase (week 2-10)
  Characterization of population pharmacokinetic parameters of orally administered BZN and BZN/E1224
Peak Plasma Concentration (Cmax) of ravuconazole and benznidazole | D0 (pre-dose), day 1 (post-dose), day 2, day 3, steady-state phase (week 2-10)
  To characterize the population pharmacokinetic parameters of orally administered BZN and BZN/E1224
Minimum Plasma Concentration (Cmin) of ravuconazole and benznidazole | D0 (pre-dose), day 1 (post-dose), day 2, day 3, steady-state phase (week 2-10)
  To characterize the population pharmacokinetic parameters of orally administered BZN and BZN/E1224
Clearance of ravuconazole and benznidazole | D0 (pre-dose), day 1 (post-dose), day 2, day 3, steady-state phase (week 2-10)
  To characterize the population pharmacokinetic parameters of orally administered BZN and BZN/E1224
Volume of Distribution of ravuconazole and benznidazole | D0 (pre-dose), day 1 (post-dose), day 2, day 3, steady-state phase (week 2-10)
  To characterize the population pharmacokinetic parameters of orally administered BZN and BZN/E1224
Plasma Terminal Half-Life (t1/2) of ravuconazole and benznidazole | D0 (pre-dose), day 1 (post-dose), day 2, day 3, steady-state phase (week 2-10)
  To characterize the population pharmacokinetic parameters of orally administered BZN and BZN/E1224

CONTACTS AND LOCATIONS:
Overall Officials: Faustino Torrico, PhD, Principal Investigator — Plataforma de Atención Integral de Pacientes con Enfermedad de Chagas. Cochabamba, Bolivia.; Joaquim Gascón, PhD, Principal Investigator — Centro de Salud Internacional, Hospital Clínico de Barcelona CRESIB - Centre de Recerca en Salut Internacional de Barcelona Barcelona, España.
Locations (3):
- Bolivia (3):
  - Plataforma de Atención Integral de Pacientes con Enfermedad de Chagas., Sucre, Chuquisaca Department
  - Plataforma de Atención Integral de Pacientes con Enfermedad de Chagas., Cochabamba
  - Plataforma de Atención Integral de Pacientes con Enfermedad de Chagas., Tarija

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saade U, de Boer J, Scandale I, Altcheh J, Pottel H, Chatelain E, Zrein M. Early assessment of antibodies decline in Chagas patients following treatment using a serological multiplex immunoassay. Nat Commun. 2024 Dec 3;15(1):10530. doi: 10.1038/s41467-024-54910-x. PMID 39627222
- [Derived] Torrico F, Gascon J, Barreira F, Blum B, Almeida IC, Alonso-Vega C, Barboza T, Bilbe G, Correia E, Garcia W, Ortiz L, Parrado R, Ramirez JC, Ribeiro I, Strub-Wourgaft N, Vaillant M, Sosa-Estani S; BENDITA study group. New regimens of benznidazole monotherapy and in combination with fosravuconazole for treatment of Chagas disease (BENDITA): a phase 2, double-blind, randomised trial. Lancet Infect Dis. 2021 Aug;21(8):1129-1140. doi: 10.1016/S1473-3099(20)30844-6. Epub 2021 Apr 6. PMID 33836161